CLINICAL TRIAL: NCT04310722
Title: Dissemination and Resistance Mechanisms of Carbapenem-resistant Gram-negative Bacilli and Methicillin-resistant Staphylococcus Aureus in Intensive Care Units in China
Brief Title: Gram-negative Bacilli and MRSA Screening in ICU in China
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sir Run Run Shaw Hospital (Other)
Collaborators: University of Birmingham (Other)
Responsible Party: Principal Investigator, Jian-cang Zhou M.D., Prof., Sir Run Run Shaw Hospital
Other Study IDs: SRRSH-DETECTIVE-CHINA
Record Dates: First submitted 2020-03-13; First posted 2020-03-17 (Actual); Last update posted 2020-03-20 (Actual); Status verified 2020-03

CONDITIONS: Infections, Bacterial
MeSH Terms: conditions — Bacterial Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The specimen will be collected from the environment and the patients in ICU setting, then the strains will be stored and DNA will be extracted.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Gram-negative bacilli and MRSA infections in ICU: Carbapenem-resistant Gram-negative bacilli [Carbapenem-resistant Acinetobacter baumannii (CRAB), Carbapenem-resistant Klebsiella pneumoniae (CRKP), and Carbapenem-resistant Pseudomonas aeruginosa (CRPsA) ] and methicillin-resistant Staphylococcus aureus (MRSA) is prevalent around the world, and the isolation rate and resistance rate has increasing in China, especially in ICU. So, investigators aim to study transmission mechanism, resistance mechanism and horizontal transfer mechanism of these pathogens.
  Interventions: Other: None intervention. This is an observational study.

INTERVENTIONS:
Other: None intervention. This is an observational study. — None intervention. This is an observational study.

SUMMARY:
Carbapenem-resistant Gram-negative bacilli [Carbapenem-resistant Acinetobacter baumannii (CRAB), Carbapenem-resistant Klebsiella pneumoniae (CRKP), and Carbapenem-resistant Pseudomonas aeruginosa (CRPsA) ] and methicillin-resistant Staphylococcus aureus (MRSA) is prevalent around the world, and the isolation rate and resistance rate has increasing in China. The limited treatment and high mortality rate of these pathogens infections has resulted in difficulty in clinical anti-infection treatment, so it is urgent to illustrate the transmission mechanism, resistance mechanism and horizontal transfer mechanism of resistance genes in intensive care unit (ICU). Furthermore, this study was aimed to investigate the epidemiology and risk factors, outcomes and the rationality of the current therapy for these pathogens infections in China.

DETAILED DESCRIPTION:
Based on the previous study, investigators plan to screen for CRKP, CRAB, CRPsA and MRSA isolates from ICU settings, medical workers and patients, and establish the CRKP, CRAB, CRPsA and MRSA genome and transcriptome database through next-generation sequencing. Under the guide of British bioinformatics and hospital-acquired infection control experts, investigators will build the transmission mechanism model of CRKP, CRAB, CRPsA and MRSA combined with the clinical data to reveal the route and rule of transmission. And the study will also demonstrate that the resistance mechanism and horizontal transfer mechanism of resistance genes of carbapenems and other main antimicrobial agents. Investigators will also set up alerting platform and new antibiotic susceptible system based on the genome and transcriptome. These results will provide scientific evidence to rational application of antimicrobial agents, reduction the prevalence of CRKP, CRAB, CRPsA and MRSA, improvement the prognosis of infections and development of new antimicrobial agents. Finally, to find the prevalence, risk factors, outcome and the rationality of the current therapy for these pathogens infections in China.

ELIGIBILITY:
Inclusion Criteria:

* Patients infected by CRAB isolated from throat swabs, rectal swabs, gastric tubes, tracheal intubations, tracheostomy tubes, and nasointestinal tubes
* Patients infected by CRKP isolated from throat swabs, rectal swabs, gastric tubes, tracheal intubations, tracheostomy tubes, and nasointestinal tubes
* Patients infected by CRPsA isolated from throat swabs, rectal swabs, gastric tubes, tracheal intubations, tracheostomy tubes, and nasointestinal tubes
* Patients infected by MRSA collected from throat swabs, rectal swabs, gastric tubes, tracheal intubations, tracheostomy tubes, and nasointestinal tubes

Exclusion Criteria:

* Mixed infections of other pathogens
* Virus infections
* Other infections caused by other pathogens, such as fungus

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients whose primary diagnosis is infections caused by CRAB, CRKP, CRPsA, or MRSA
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-08-06 (Actual); Primary Completion 2020-10 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Microbiological infection diagnosis | Through study completion, up to one year
  1. Culture positive results confirmed the infection of CRAB, CRKP, CRPsA and MRSA
  2. 8 participants will collect the samples from the patients and environment in one ICU and isolation rate of CRAB, CRKP, CRPsA and MRSA will be obtained
  3. Molecular characteristics of CRAB, CRKP, CRPsA and MRSA using multilocus sequence type (MLST), pulsed field gel electrophoresis (PFGE) and whole-genome sequencing (WGS)

CONTACTS AND LOCATIONS:
Overall Officials: Yun-song Yu, Dr., Principal Investigator — Zhejiang University
Locations (1):
- Sir Run Run Shaw Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided